CLINICAL TRIAL: NCT06605456
Title: The Effect of Proprioceptive Neuromuscular Facilitation Combined With Postural Education on Pressure Pain Threshold in Upper Back Among Students With Upper Cross Syndrome: an Experimental Study
Brief Title: Proprioceptive Neuromuscular Facilitation Combined With Postural Education in Upper Cross Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gulf Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB/COHS/STD/16/FEB-2023
Record Dates: First submitted 2024-09-18; First posted 2024-09-20 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Upper Cross Syndrome
Keywords: Upper cross syndrome; Postural correction; Neck pain; Upper back pain; Neuromuscular facilitation
MeSH Terms: conditions — Oculocerebral hypopigmentation syndrome type Preus; Neck Pain; Back Pain | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Intervention Model Description: Group A, who were assigned the PNF neck pattern intervention, a rhythmic initiation technique was implemented.
  Group B were assigned active neck muscle stretching as well as self-isometric strengthening exercises, targeting all cervical muscle groups.
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor was blinded to the randomization of subjects into the intervention groups
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: PNF with postural education (Experimental): PNF neck pattern intervention with a rhythmic initiation technique implemented. This exercise intervention consisted of a two-phase exercise set: stretching the muscles and strengthening them
  Interventions: Other: Proprioceptive neuromuscular facilitation with postural education
- Group B: Active neck muscle stretching and strengthening exercises (Active Comparator): Active neck muscle stretching and self-isometric strengthening exercises, targeting all cervical muscle groups.
  Interventions: Other: Active neck muscle stretching and strengthening exercises

INTERVENTIONS:
Other: Proprioceptive neuromuscular facilitation with postural education — Phase 1: Active Rhythmic Initiation The exercise was demonstrated to the students in a seated position, as sitting is considered the functional position for neck motion and stability. Then, the exercises was passively practiced on the students using tactile input. After passive demonstration, students were asked to perform the same exercise actively and verbal commands were used to guide and correct them.
  Phase 2: Resisted Rhythmic Initiation "Modified" The investigators applied resistance by placing the palm of one hand on the right side of the chin to strengthen the muscles. Then, resisted scapular posterior depression PNF exercise also employed.
  Also received a comprehensive postural education program to emphasize the importance of proper posture. The program was divided into three sections, which focused on the effects of good and bad posture, as well as practical demonstration.
  Arms: Group A: PNF with postural education
Other: Active neck muscle stretching and strengthening exercises — Phase 1: Active Muscle Stretching In this phase, participants were instructed on performing active muscle stretching exercises for all cervical muscles, including neck flexors, extensors, lateral flexors and neck rotators. Each stretch was held for a period of 25-30 seconds and repeated three times.
  Phase 2: Self-Isometric Strengthening Participants were provided with a demonstration of self-isometric strengthening exercise for the neck muscles. The exercises involved six movement patterns: cervical flexion, cervical extension, right/left lateral flexion and right/left rotation. For each exercise the participants were required to apply resistance against the direction of movement using their hand without allowing any motion in the neck.
  Also received a comprehensive postural education program to emphasize the importance of proper posture. The program was divided into three sections, which focused on the effects of good and bad posture, as well as practical demonstration.
  Arms: Group B: Active neck muscle stretching and strengthening exercises

SUMMARY:
The aim of this study was to investigate the effectiveness of PNF and conventional neck stretching, combined with a postural education program in improving forward head posture in students with clinical signs and symptoms of UCS. The study included a sample of undergraduate Gulf Medical University students with clinical signs and symptoms of UCS. A total of 24 samples were divided into two groups of 12. Group A received PNF pattern neck stretching and self-resisted neck PNF pattern, whereas Group B received Conventional neck stretches along with isometric strengthening of the neck muscles. Both groups were given a common postural education program. The intervention duration was 5 days per week for 4 weeks.

DETAILED DESCRIPTION:
Collegiate students are prone to adopt slouched posture and develop muscular imbalance which is considered as a causative factor for the development of UCS. Studies have shown that students in medical universities have a higher risk of developing UCS. Even though PNF is considered to be simple and effective to improve inter and intramuscular coordination, its application to collegiate students with UCS is limited. Application of PNF combined with postural education programs may benefit the students to reduce UCS-associated clinical problems such as reduced forward head posture, pain intensity and improving muscle strength etc. Our current study might open the door of simple and effective management of UCS among collegiate students. Therefore, our study was conducted to find out the effect of PNF and active muscle stretching, both in combination with postural education programs, on forward head posture of the students with upper crossed syndrome.

Objectives:

● To compare the effect of PNF with active muscle stretching, both in combination with postural education programs on forward head posture of students with upper cross syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Students of Gulf Medical University.
* Both genders.
* Age between 18 - 30 years.
* Presence of clinical signs and symptoms of UCS.
* Presence of FHP with CVA of 49 degrees and below.

Exclusion Criteria:

* Musculoskeletal disorder such as strain, sprain, scoliosis.
* Students participating in any other interventions.
* Nutritional deficiencies.
* Unwilling participate.
* Degenerative joint disorder
* Neurologically unstable individuals

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2023-02-16 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-07-15 (Actual)

PRIMARY OUTCOMES:
Forward Head Posture | Day one before the treatment, Four weeks post treatment.
  Measured by using a mobile phone app (physio master) and have taken craniovertebral angle, sagittal head tilt, and, head shoulder angle to identify a forward head posture.

SECONDARY OUTCOMES:
Trigger point tenderness | Day one before the treatment, Four weeks post treatment.
  The manual palpation method was applied to specific muscle groups associated with UCS, including the upper trapezius, rhomboids, levator scapulae, and sternomastoid (STM). The grading scale involved four grades: grade 1, where the patient complains of pain; grade 2, where the patient winces on palpation; grade 3, where the patient withdraws from palpation; and grade 4, where the patient is not allowed to be touched.
Cervical spine range of motion | Day one before the treatment, Four weeks post treatment.
  To assess the range of motion (ROM) of the cervical muscle groups, an Acumar single & Dual inclinometer (Lafayette instrument, models ACU001 & ACU002) was utilized. For neck flexion, the inclinometer was placed on the top of the student's head, and the other end of the inclinometer was positioned on the T1 vertebra while the student was seated. The same method was applied for measuring neck extension and left/right lateral flexion. To measure left/right rotation, the participants were asked to be in a supine position, and the inclinometer was placed on the forehead as the main reference point. During each measurement, three trials were conducted, and the mean value of the three trials was calculated to determine the ROM for each specific movement.

CONTACTS AND LOCATIONS:
Overall Officials: Ramprasad Muthukrishnan, PhD, Study Chair — Gulf Medical University
Locations (1):
- Gulf Medical University, Al Jurf, Ajman Emirate, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No
Data might be shared based on the request